CLINICAL TRIAL: NCT04348773
Title: Assessment of Tooth Shade After De- and Re-Hydration During Clinical Restorative Procedures (A Randomized Clinical Trial)
Brief Title: Assessment of Tooth Shade After De- and Re-Hydration During Clinical Restorative Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Abou-steit, Sameh Abou-Steit, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-2020-4-040
Record Dates: First submitted 2020-04-09; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Tooth Shade
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dehydration (Experimental)
  Interventions: Procedure: Dehydration
- Rehydration (Experimental)
  Interventions: Procedure: Rehydration

INTERVENTIONS:
Procedure: Dehydration — Dehydration of the natural tooth by tooth isolation
  Arms: Dehydration
Procedure: Rehydration — Rehydration
  Arms: Rehydration

SUMMARY:
The aim of this study was to investigate any change in tooth color resulting from dehydration resulted from rubber dam application and the time required for any change to return to baseline and to investigate the nature of change and areas of the teeth most affected.

DETAILED DESCRIPTION:
Architecturally speaking, a smile comprises 60% of the weight of our face. Subconsciously, a smile has a visual impact on people appearance. Also statistically reveal that people place a high value on their smiles according to the American academy of cosmetic dentistry survey (AACD)2017. As the population becomes increasingly aware of the role teeth play in appearance, patients' expectations of aesthetics in contemporary dentistry are ever increasing. So practicing esthetic dentistry that is defined as reproducing natural looking teeth by creating perfect esthetic restorations has been for long time a strict challenge due to many materials' limitations impacting either shade integration or surface quality, and possibly colour stability.

Tooth colour was the main reason for patient dissatisfaction in a survey concerned with esthetic appearance.(1) Thus accurate shade measurement together with proper communication of tooth colour is integral to a successful aesthetic outcome.(2) It is compulsory that clinicians understand the light interaction with tooth structures as well as the proper histo-anatomic principles for a better material and shade selection during direct and indirect restorative procedures. Tooth structures form a complex optical medium for light as it passes through enamel, dentino-enamel complex and dentin in terms of gradient between transparency (complete transmission of light) and opacification (complete reflection of light).(3)Furthermore, this behavior changes over the years, as tissues change in morphology and composition. Comprehension of dynamic aging of tooth structures is a key for success when selecting the proper value and chromaticity for restorative materials.(4,5) Thus clinicians and technicians should have sufficient training in tooth shade selection. For achieving excellent esthetic outcomes there are four main contributing variables: Dynamic Light Interaction, Histo-anatomical Features, Smilography and the 9 Elements of visual synthesis.(3) In the modern dental practice, restoring the optical features of the intact tooth presents a challenging task, due to the inherent translucent nature of enamel, the dentinoenamel complex (DEC) and dentin. Translucent materials offer a significant color measurement challenge since they interact with light in a far more complex manner than most other materials. The old traditional visual estimation approaches that solely employ the Munsell color model system based on hue, chroma, and value (H/C/V) dominating the dental market appear to be insufficient when assigning the relevant information among the dental team members (clinician/technician/patient).(6) In 1931 The Commission Internationale de l'Eclairage (CIE) defined a standard light source, developed a standard observer and enabled the calculation of tri-stimulus x, y, z values, which represent how the human visual system responds to a given colour and allows us to transform spectral energy data into meaningful colour data. It should be noted that the DE in the L*a*b* colour space indicates the degree of colour difference not the direction of the colour difference. It is frequently interpreted in dental literature that a DE of 1 is the 50:50 perceptibility threshold. The hues of natural teeth tend to be in the yellow to yelloworange range, determined mainly by the colour of dentine, with enamel playing only a minor role through scattering at wavelengths in the blue range.(7) Instruments for clinical shade matching include spectrophotometers, colourimeters and digital imaging systems.(8) It has been reported that VITA Easyshade has to be the most reliable instrument in both in vitro and in vivo circumstances.(2) It has been reported that dehydration of teeth can make them appear whiter by increasing enamel opacity when examined by The Easyshade as the light can no longer scatter from hydroxyapatite crystal to crystal.(6,10,11)The resulted loss of translucency on dehydration therefore causes more reflection masking the color of the underlying dentine and thus appears lighter. Russell et al.(12) applied a rubber dam to the anterior teeth of seven subjects and allowed the teeth to dehydrate for 15 min that was measured using a spectrophotometer and further three spectrophotometric measurements were taken at 10 min intervals after removal of rubber dam and tooth rehydration. It was noticed that tooth colour had become lighter and less saturated after dehydration and the colour of the teeth returned to their baseline values 20 min after removal of the rubber dam. Most dental procedures cause some dehydration of teeth.(13-16) It is recommended to record the shade of teeth at the begining of the appointment but there is insufficient evidence in the dental literature to support it.(14) Color mismatch between restoration and natural teeth is a common complaint resulting in remake of restorations and increased expense.(2) As most dental procedures lead to dehydration of teeth which can alter their shade and may lead to errors in shade matching. And in order to avoid unacceptable mismatch of color between natural teeth and dental restoration, it is important that the shade matching procedure is carried out at the beginning of the appointment. Thus the aim of this study was to investigate any change in tooth color resulting from dehydration resulted from rubber dam application and the time required for any change to return to baseline and to investigate the nature of change and areas of the teeth most affected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unrestored intact maxillary central incisors with no tooth bleaching performed during the previous year.

Exclusion Criteria:

* Presence of any restorations or fixed orthodontic appliance or any fixed retainers on central incisors

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical spectrophotometric assessment of tooth shade change | 10, 30, 40 and 60 minutes
  Using Easyshade V clinical spectrophotometer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Zohairy, PhD, Study Director — Head of Operative department
Locations (1):
- Faculty of Dentistry, Cairo Univerity, Cairo, Egypt

REFERENCES:
- [Background] Samorodnitzky-Naveh GR, Geiger SB, Levin L. Patients' satisfaction with dental esthetics. J Am Dent Assoc. 2007 Jun;138(6):805-8. doi: 10.14219/jada.archive.2007.0269. PMID 17545270
- [Background] Burki Z, Watkins S, Wilson R, Fenlon M. A randomised controlled trial to investigate the effects of dehydration on tooth colour. J Dent. 2013 Mar;41(3):250-7. doi: 10.1016/j.jdent.2012.11.009. Epub 2012 Nov 14. PMID 23160038
- [Background] Bazos P, Magne P. Bio-Emulation: biomimetically emulating nature utilizing a histoanatomic approach; visual synthesis. Int J Esthet Dent. 2014 Autumn;9(3):330-52. PMID 25126615
- [Background] Hariri I, Sadr A, Nakashima S, Shimada Y, Tagami J, Sumi Y. Estimation of the enamel and dentin mineral content from the refractive index. Caries Res. 2013;47(1):18-26. doi: 10.1159/000342416. Epub 2012 Oct 10. PMID 23051596
- [Background] Hariri I, Sadr A, Shimada Y, Tagami J, Sumi Y. Effects of structural orientation of enamel and dentine on light attenuation and local refractive index: an optical coherence tomography study. J Dent. 2012 May;40(5):387-96. doi: 10.1016/j.jdent.2012.01.017. Epub 2012 Feb 7. PMID 22342164
- [Background] Joiner A. Tooth colour: a review of the literature. J Dent. 2004;32 Suppl 1:3-12. doi: 10.1016/j.jdent.2003.10.013. PMID 14738829
- [Background] Paul S, Peter A, Pietrobon N, Hammerle CH. Visual and spectrophotometric shade analysis of human teeth. J Dent Res. 2002 Aug;81(8):578-82. doi: 10.1177/154405910208100815. PMID 12147751
- [Background] Brewer JD, Wee A, Seghi R. Advances in color matching. Dent Clin North Am. 2004 Apr;48(2):v, 341-58. doi: 10.1016/j.cden.2004.01.004. PMID 15172604
- [Background] Douglas RD, Steinhauer TJ, Wee AG. Intraoral determination of the tolerance of dentists for perceptibility and acceptability of shade mismatch. J Prosthet Dent. 2007 Apr;97(4):200-8. doi: 10.1016/j.prosdent.2007.02.012. PMID 17499089
- [Background] Stevenson B. Current methods of shade matching in dentistry: a review of the supporting literature. Dent Update. 2009 Jun;36(5):270-2, 274-6. doi: 10.12968/denu.2009.36.5.270. PMID 19585849
- [Background] Dozic A, Kleverlaan CJ, El-Zohairy A, Feilzer AJ, Khashayar G. Performance of five commercially available tooth color-measuring devices. J Prosthodont. 2007 Mar-Apr;16(2):93-100. doi: 10.1111/j.1532-849X.2007.00163.x. PMID 17362418
- [Background] Russell MD, Gulfraz M, Moss BW. In vivo measurement of colour changes in natural teeth. J Oral Rehabil. 2000 Sep;27(9):786-92. doi: 10.1046/j.1365-2842.2000.00610.x. PMID 11012854
- [Background] Meng Z, Yao XS, Yao H, Liang Y, Liu T, Li Y, Wang G, Lan S. Measurement of the refractive index of human teeth by optical coherence tomography. J Biomed Opt. 2009 May-Jun;14(3):034010. doi: 10.1117/1.3130322. PMID 19566303
- [Background] Suliman S, Sulaiman TA, Olafsson VG, Delgado AJ, Donovan TE, Heymann HO. Effect of time on tooth dehydration and rehydration. J Esthet Restor Dent. 2019 Mar;31(2):118-123. doi: 10.1111/jerd.12461. Epub 2019 Feb 23. PMID 30801926